CLINICAL TRIAL: NCT03600311
Title: Using Resistance Exercise and Protein Consumption to Protect Bone Health During Weight Loss
Brief Title: Resistance Exercise and Protein During Weight Loss
Acronym: RIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17933
Record Dates: First submitted 2018-07-09; First posted 2018-07-26 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Weight Loss; Starvation
MeSH Terms: conditions — Weight Loss; Starvation | interventions — Caloric Restriction; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Energy Balance (Placebo Comparator): Participants will be in energy balance and consume 1.2 g/kg BW protein. They will be provided 30 g of maltodextrin following exercise.
  Interventions: Other: Energy Balance; Dietary Supplement: Post-Exercise Carbohydrate; Dietary Supplement: Calcium and Vitamin D
- Caloric Restriction and CHO Supp (Active Comparator): Participants will be calorie restricted to 15 kcal/kg FFM/day and consume 1.2 g/kg BW protein. They will be provided 30 g of maltodextrin following exercise.
  Interventions: Other: Caloric Restriction; Dietary Supplement: Post-Exercise Carbohydrate; Dietary Supplement: Calcium and Vitamin D
- Caloric Restriction and PRO Supp (Experimental): Participants will be calorie restricted to 15 kcal/kg FFM/day and consume 1.2 g/kg BW protein. They will be provided 30 g of whey protein following exercise.
  Interventions: Other: Caloric Restriction; Dietary Supplement: Post-Exercise Protein; Dietary Supplement: Calcium and Vitamin D

INTERVENTIONS:
Other: Caloric Restriction — Participants will consume 15 kcal/kg FFM/day.
  Arms: Caloric Restriction and CHO Supp; Caloric Restriction and PRO Supp
Dietary Supplement: Post-Exercise Protein — Participants will ingest 30 g of protein following exercise.
  Arms: Caloric Restriction and PRO Supp
Other: Energy Balance — Participants will consume 40 kcal/kg FFM/day.
  Arms: Energy Balance
Dietary Supplement: Post-Exercise Carbohydrate — Participants will ingest 30 g of carbohydrate following exercise.
  Arms: Caloric Restriction and CHO Supp; Energy Balance
Dietary Supplement: Calcium and Vitamin D — Participants will be supplied Calcium and Vitamin D supplements throughout the study period matched to the CON condition.

SUMMARY:
The purpose of this study is to determine if post-exercise protein supplementation can rescue the anabolic response of muscle and bone to resistance exercise during caloric restriction.

DETAILED DESCRIPTION:
1. Preliminary Testing Prior to the study start, participants will be weighed and body composition will be determined using bioimpedance analysis. Then participants will undergo a 5RM barbell back squat exercise testing procedure.
2. Randomization

   Participants will proceed through each of the following conditions lasting 3 days:

   CON: Participants will be in energy balance and consume 1.2 g protein/kg BW/day. Participants will be provided 30 g maltodextrin post-exercise.

   CR+C: Participants will be restricted to 15 kcal/kg FFM/day and consume 1.2 g protein/kg BW/day. Participants will be provided 30 g maltodextrin post-exercise.

   CR+P: Participants will be restricted to 15 kcal/kg FFM/day and consume 1.2 g protein/kg BW/day. Participants will be provided 30 g whey protein post-exercise.
3. Diet Prescription Dietary energy intake will be controlled using clinical products, maltodextrin and whey protein isolate to meet target energy intakes. Participants will receive calcium and Vitamin D supplementation throughout the study.
4. Exercise Prescription Participants will perform one bout of 5 sets of 5 repetitions of barbell back squat exercise on the morning of Day 3 each condition. Additional exercise and intense physical activity will be prohibited.
5. Assessments Body weight and composition (DXA + BIA), fasting blood draws for assessment of metabolic and anabolic hormones and questionnaires will be conducted before and after each condition. A 24-hour serial blood draw procedure will be conducted following each workout session on each Day 3.
6. Washout Once a participant completes a study condition, participants will continue to take daily body weights at home for up to one week. Then participants will be required to wait one more week before completing their next condition during which they will resume regular diet and physical activity.

ELIGIBILITY:
Baseline Inclusion Criteria:

* Weigh at least 110 lbs
* Weight-Stable (2.5 kg) within the past six months
* Height-Stable (< 0.25 inches) within the past year
* 3 years of resistance training experience

Tested Inclusion Criteria:

- <20% body fat (men) or <30% body fat (women)

Exclusion Criteria:

* Lactose intolerant
* Pregnancy
* Taking interfering medications such as steroids, thyroid or growth hormones

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Serum [IGF-1] (ng/mL) | Baseline, Pre-Exercise, 0-24 Hours Post-Exercise
  Measured via ELISA
Change in Serum [GH] (pg/mL) | Baseline, Pre-Exercise, 0-24 Hours Post-Exercise
  Measured via ELISA
Change in Serum [IGFBP-3] (ng/mL) | Baseline, Pre-Exercise, 0-24 Hours Post-Exercise
  Measured via ELISA
Change in Serum [P1NP] (pg/mL) | Baseline, Pre-Exercise, 0-24 Hours Post-Exercise
  Measured via ELISA
Change in Serum [CTX] (ng/mL) | Baseline, Pre-Exercise, 0-24 Hours Post-Exercise
  Measured via ELISA
Change in Serum [Sclerostin] (pmol/L) | Baseline, Pre-Exercise, 0-24 Hours Post-Exercise
  Measured via ELISA

SECONDARY OUTCOMES:
Change in Body Weight (kg) | Baseline and Day 4
  Measured via Stadiometer
Change in Body Fat Percentage (%) | Baseline and Day 4
  Measured via DXA and BIA
Change in Perceived Hunger (mm or %) | Baseline and Day 4
  Measured on Visual Analog Scale within Survey

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Koehler, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- Sports and Exercise Nutrition Laboratory, Department of Nutrition and Health Sciences, Ruth Leverton Hall, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No